CLINICAL TRIAL: NCT00320164
Title: Anti-Pseudomonas Immune Status and Dendritic Cell Preparation in Normal Individuals
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: Dendritic Cells
Record Dates: First submitted 2006-04-27; First posted 2006-05-03 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Healthy
Keywords: Healthy Volunteers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Leukapheresis: Subject's peripheral blood mononuclear cells are collected via leukapheresis.
- Group B: Buffy Coats Collection: Subject's peripheral blood mononuclear cells are collected via the buffy coats from blood.

SUMMARY:
This protocol aims to collect human peripheral blood mononuclear cells for the production of dendritic cells (DC). There are two ways to collect human peripheral blood mononuclear cells in this protocol. One is by using the method of leukapheresis from normal healthy adults. The other is by drawing the blood from normal healthy adults and then getting the buffy coats from the blood.

DETAILED DESCRIPTION:
One objective of these studies on DC is to complete a preclinical development for a human study of a candidate anti-Pseudomonas aeruginosa vaccine consisting of autologous dendritic cells primed with heat-inactivated P. aeruginosa (PA) strain POA1 and expressing the T-cell costimulatory molecule CD40 ligand (CD40L). The other objective is to complete a preclinical development for a human study of a candidate anti-anthrax vaccine. Prior to testing the vaccine in humans, the Food and Drug Administration will require preclinical and Good Manufacturing Practice (GMP) practice batches of dendritic cells. The intent of the leukapheresis or collecting the buffy coats is to provide the biological materials for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* All study subjects must be capable of providing informed consent.
* Normal male or female, age 18 and older.
* Not taking corticosteroids
* Not taking any prescription or over-the-counter medication, except acetaminophen (tylenol)
* Participants of Group A must have adequate peripheral veins for leukapheresis
* Study subjects should not be taking experimental medications.
* Females cannot be pregnant.

Exclusion Criteria:

* Individuals who do not meet the inclusion criteria will be unable to participate in the protocol.
* Individuals with active infection in the 3 weeks prior to beginning the protocol will not be able to participate.
* Individuals with evidence of significant cardiac, pulmonary, renal, endocrine, central nervous system, major psychiatric disorder that would prevent compliance or substance abuse, musculoskeletal disease or immunodeficiency disease, (including evidence of human immunodeficiency virus infection, HIV) will be unable to participate in the protocol.
* Individuals participating in any other experimental clinical studies.
* Women who are pregnant or nursing.
* Active or recent drug users

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group A is for leukapheresis and Group B is for buffy coats collection. We will use either Group A or Group B or both to collect mononuclear cells. The source of potential subjects in both groups will be normal individuals recruited from the population of healthy individuals. Accrual will be random with no bias as to gender or racial/ethnic group. Nevertheless, because the accrual process will be random, it is possible that there may be differences in the proportion of males and females, and racial/ethnic groups. The study volunteers will be recruited through IRB approved advertisements placed in local newspapers and fliers. All efforts will be made to recruit women and minorities.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil R. Hackett, Ph.D., Principal Investigator — Weill Medical College of Cornell University

IPD SHARING:
Plan to Share IPD: Undecided